CLINICAL TRIAL: NCT00321958
Title: Cryotherapy Ablation of Barrett's Esophagus and Early Esophageal Cancer
Brief Title: Study of Cryotherapy Treatment of Barrett's Esophagus and Early Esophageal Cancer
Status: Terminated | Type: Observational
Why Stopped: The sponsor determined that adequate data had been acquired.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: CSA Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Bruce Greenwald, PI, University of Maryland, Baltimore
Other Study IDs: H-27406; CCT Number = 3511 (Other Grant/Funding Number: UMB)
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Barrett Esophagus; Esophageal Neoplasms; Deglutition Disorders; GERD; Neoplasm
Keywords: Barrett Esophagus; Esophageal Neoplasm; Deglutition disorders; Cryotherapy; Cryosurgery; GERD; Neoplasm; Esophagus; Endoscopy, Digestive System
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Deglutition Disorders; Gastroesophageal Reflux; Neoplasms | interventions — Cryoelectron Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CSA System (CryoSpray AblationTM System) — 10 second spray times
  Other Names: CSA; Cryo
Device: CryoSpray Ablation — 10 second spray times
  Other Names: CSA; cryo

SUMMARY:
The purpose of this study is to confirm the effectiveness and safety of a new medical device which sprays liquid nitrogen through an upper endoscope (cryotherapy) to treat Barrett's esophagus with high-grade dysplasia and early esophageal cancer. It is hypothesized that this treatment will remove the abnormal lining of the esophagus and allow the normal esophageal lining to return.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) with high grade dysplasia (HGD) is a precursor of esophageal adenocarcinoma. Eliminating this condition may control the current rapid rise of adenocarcinoma. Ablative techniques are attempted to avoid the high morbidity and mortality of esophagectomy or for use in patients who cannot undergo surgery. Current ablative techniques have achieved mucosal ablation with variable success but are associated with high cost, patient discomfort and/or significant complications. A novel device which sprays liquid nitrogen through an upper endoscope (cryotherapy) has been shown to be a safe and effective procedure to ablate the esophageal mucosa in swine and dog models and in pilot studies in humans. Successful reversal of BE, LGD, HGD and superficial adenocarcinoma and squamous cell carcinoma have been demonstrated when cryotherapy with this device is followed by healing of the esophageal lining in a low acid environment.

This study is undertaken to demonstrate the efficacy and safety in the ablation of Barrett's esophagus with high-grade, neoplasia, and severe esophageal squamous dysplasia and to confirm preliminary results in humans.

ELIGIBILITY:
Inclusion Criteria:

* High Grade-IMCancer:

  * Diagnosis of Barrett's esophagus and high-grade dysplasia or intramucosal carcinoma
  * Deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney or liver disease; or refusal of surgical intervention after a thorough discussion of the highly experimental nature of cryotherapy
  * CT scan of the chest and abdomen with oral and intravenous contrast (unless allergic), demonstrating no evidence of advanced esophageal cancer (extension into or through the wall or lymph node involvement)
  * Endoscopic ultrasound evaluation demonstrating no evidence of metastatic lymph node involvement or extension of carcinoma beyond the mucosa
  * Pathology review of esophageal biopsies by two independent reviewers, including at least one from the Department of Pathology at the University of Maryland, to confirm the diagnosis of Barrett's esophagus with HGD and/or IMCA
  * Presentation and discussion at Thoracic Tumor Board
* Mucosal/submucosal cancer:

  * Diagnosis of esophageal carcinoma
  * Deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney or liver disease; or refusal of surgical intervention after a thorough discussion of the highly experimental nature of cryotherapy
  * CT scan of the chest and abdomen with oral and intravenous contrast (unless allergic), demonstrating no evidence of advanced esophageal cancer (extension through the wall or lymph node involvement)
  * Endoscopic ultrasound evaluation demonstrating no evidence of metastatic lymph node involvement and primary lesion extending into submucosa or muscularis propria (T1smN0 or T2N0)
  * Presentation and discussion at Thoracic Tumor Board
  * Patients who have undergone previous ablation therapies are eligible for this study.
* Severe squamous dysplasia:

  * Diagnosis of severe dysplasia within esophageal squamous mucosa
  * Deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney or liver disease; or refusal of surgical intervention after a thorough discussion of the highly experimental nature of cryotherapy
  * CT scan of the chest and abdomen with oral and intravenous contrast (unless allergic), demonstrating no evidence of advanced esophageal cancer (extension into or through the wall or lymph node involvement)
  * Endoscopic ultrasound evaluation demonstrating no evidence of metastatic lymph node involvement or extension of carcinoma beyond the mucosa
  * Pathology review of esophageal biopsies by two independent reviewers, including at least one from the Department of Pathology at the University of Maryland, to confirm the diagnosis
  * Presentation and discussion at Thoracic Tumor Board

Exclusion Criteria:

* Age less than 18 years
* Co-morbid illness expected to cause death within 6 months
* Pregnancy
* Medically unfit or other contraindication to tolerate upper endoscopy
* Inability to tolerate therapy with a proton pump inhibitor (PPI)
* Refusal or inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have Barrett's esophagus and high grade dysplasia or intramucosal cancer, squamous dysplasia, or mucosal/submucosal cancer
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
HGD or inoperable intramucosal or submucosal carcinoma and severe squamous dysplasia: measure of reduction in size of HGD or carcinoma | Study end
  HGD or inoperable intramucosal or submucosal carcinoma and severe squamous dysplasia: measure of reduction in size of HGD or carcinoma

SECONDARY OUTCOMES:
HGD or inoperable intramucosal carcinoma: Rate of complete ablation of all BE and associated HGD or intramucosal carcinoma | Study midpoint and end
  HGD or inoperable intramucosal carcinoma: Rate of complete ablation of all BE and associated HGD or intramucosal carcinoma
Number of treatment sessions needed to ablate BE and associated HGD or intramucosal carcinoma | Study end
  Number of treatment sessions needed to ablate BE and associated HGD or intramucosal carcinoma
Rate of adverse events | Throughout study
  Rate of adverse events
Inoperable mucosal or submucosal carcinoma (T1mN0, T1smN0 and T2N0): Time to cancer recurrence | Throughout study
  Inoperable mucosal or submucosal carcinoma (T1mN0, T1smN0 and T2N0): Time to cancer recurrence
Inoperable severe squamous dysplasia: Rate of complete ablation of all dysplasia | Study end
  Inoperable severe squamous dysplasia: Rate of complete ablation of all dysplasia
Number of treatment sessions needed to ablate dysplasia | Throughout study
  Number of treatment sessions needed to ablate dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Greenwald, M.D., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland School of Medicine and Greenebaum Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Johnston, M.H. Endoscopic cryotherapy: A new ice age in gastroenterology? [Electronic version]. Medscape Gastroenterology 2:(4)2000.
- [Background] Johnston, M.H., Eastone, J.A., & Horwhat, J.D. Reversal of Barrett's esophagus with cryotherapy [Abstract]. American Journal of Gastroenterology 98: (9,Suppl), A30,S11, 2003.
- [Background] Johnston, M., Horwhat, J., Dubois, A., & Schoenfeld, P. Endoscopic cryotherapy in the swine esophagus: A follow-up study [Abstract]. Gastrointestinal Endoscopy 49: AB126, 1999.
- [Background] Johnston, M.H., Horwhat, J.D., Haluska, O., & Moses, F.M. Depth of injury following endoscopic spray cryotherapy: EUS assisted evaluation of mucosal ablation and subsequent healing in the swine model [Abstract] [Electronic version]. Gastrointestinal Endoscopy 51: AB98,3462, 2000.
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Johnston, M.H., Schoenfeld, P., Mysore, J., Kita, J.A., & Dubois, A. Endoscopic cryotherapy: A new technique for tissue ablation in the esophagus [Abstract]. American Journal of Gastroenterology 92: A44, 1997.
- [Background] Eastone, J.A., Horwhat, D., Haluska, O., Mathews, J., & Johnston, M. Cryoablation of swine esophageal mucosa: A direct comparison to argon plasma coagulation (APC) and multipolar electrocoagulation (MPEC) [Abstract] [Electronic version]. Gastrointestinal Endoscopy 53: A3448, 2001.